CLINICAL TRIAL: NCT00168922
Title: Phase II Study to Determine the Efficacy of Bendamustin (Ribomustin) in Patients With Recurrent Small Cell Bronchial Carcinoma After Cytostatic Polychemotherapy
Brief Title: Study to Determine the Efficacy of Bendamustin in Patients With Recurrent Small Cell Lung Cancer (SCLC)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: ribosepharm GmbH (Unknown)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Haema CBF SCLC UK/AS 02
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2006-04-27 (Estimated); Status verified 2001-01

CONDITIONS: Recurrent Small Cell Lung Cancer
Keywords: recurrent SCLC
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Bendamustine Hydrochloride

INTERVENTIONS:
Drug: Bendamustin/Ribomustin

SUMMARY:
Determination of response rate Assessment of toxicity and determination of "time to progression"

DETAILED DESCRIPTION:
Phase II Study to determine the efficacy of Bendamustin(Ribomustin) in patients with recurrent small cell bronchial carcinoma after cytostatic polychemotherapy

ELIGIBILITY:
Inclusion Criteria:

* Patients with histological proven, curative non treatable small lung cell carcinoma
* Recurrence >8 weeks, > 1 year after 1st line treatment with platin- and etoposide polychemotherapy, without brain metastases

Exclusion Criteria:

* Brain metastases
* WHO-PS 3 - 4

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2001-02; Study Completion 2006-12

PRIMARY OUTCOMES:
Determination of response rate ( CR + PR) after cytostatic therapy with Bendamustin 120mg/m2, day 1+2, repeat d 22
(primary goal)

SECONDARY OUTCOMES:
Assessment of toxicity, determination of time to progression, for median survival and one-year survival rate,investigation of life quality (secondary goal)

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Keilholz, MD, Principal Investigator — Charité Campus Benjamin Franklin University Clinic
Locations (1):
- Hematology & Oncology Charité CBF Berlin, Germany, Berlin, State of Berlin, Germany